

### Imperial College London

Research Governance and Integrity Team

# Consent Form for Participants Able to Give Consent

Centre name (if applicable): Study Protocol number: IRAS project ID: 326995

**Full Title of Project:** RAPPER – Relating Abdominal complications with Peritoneal Pressure Estimation and Reporting

Name of Principal Investigator:

Please initial box

#### Add/delete/amend clauses as appropriate]

| 1. | I confirm that I have read and understand the participant information sheet version |
|---|---|
| 2. | I understand that my participation is voluntary, and I am free to withdraw at any time, without giving any reason and without my legal rights nor treatment / healthcare being affected. |
| 3. | I understand that sections of any of my medical notes may be looked at by responsible individuals from NHS Trust or from regulatory authorities where it is relevant to my taking part in this research. |
| 4. | I give/do not give (delete as applicable) consent for information collected about me to be used to support other research or in the development of a new test, medication, medical device or treatment (delete as applicable) by an academic institution or commercial company in the future, including those outside of the United Kingdom (which Imperial has ensured will keep this information secure). |
| 5. | I understand that tissue samples and / or data collected from<br>me are a gift donated to Imperial College and that I will not<br>personally benefit financially if this research leads to an<br>invention and/or the successful development of a new test,<br>medication treatment, product or service. |



# Imperial College London

## Research Governance and Integrity Team

| <ol> <li>I consent to take part in (RAPPER Study: Investigating the<br/>Relationship Between Estimated Intraperitoneal Pressure and<br/>Non-Infectious PD-Related Abdominal Complications).</li> </ol> | | |
|---|---|---|
| • • | • | |
| Signature | Date | |
| Signature | Date | |
| | etimated Intraperitone ed Abdominal Compli e/mark as applicable e possibility to take p Signature | stimated Intraperitoneal Pressure and ed Abdominal Complications). e/mark as applicable) consent to e possibility to take part in other Signature Date |

1 copy for participant; 1 copy for Principal Investigator 1 copy for hospital notes

To ensure confidence in the process and minimise risk of loss, all consent forms must be printed, presented and stored in double sided format